CLINICAL TRIAL: NCT06515795
Title: Evaluation of the Safety and Efficacy of Two Isometric Exercises in the Reduction of the Blood Pressure in People With Resistant Hypertension
Brief Title: Evaluation of Two Isometric Exercises in the Reduction of the Blood Pressure in People With Resistant Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Principal Investigator, José Luís Silva Lopes, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IHGvsIWSinResistantHT
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Resistant Hypertension
Keywords: resistant hypertension; isometric exercise; handgrip; wall squat; blood pressure
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Session (No Intervention): Each participant will remain in a seated position, resting, for 40 minutes.
- Isometric Handgrip Session (Experimental): After remain in a seated position, resting, for 15 minutes, each participant will perform 4 repetitions of 2 minutes, alternating hands, maintaining the handgrip at a strength value of 30% of the maximal voluntary contraction (MVC) obtained in the initial test, with 1 minute of rest between each repetition. The exercise will be performed in a seated position. Participants will be encouraged to breathe normally and avoid the Valsalva maneuver.
  Interventions: Other: Isometric exercise
- Isometric Wall Squat Session (Experimental): After remain in a seated position, resting, for 15 minutes, each participant will perform 4 repetitions of 2 minutes, maintaining the squat position with their back against the wall, with 2 minutes of rest (in a seated position) between each repetition. The knee joint angle will be defined using a fixed goniometer attached with Velcro to the thigh and leg. This angle corresponds to the knee position at 95% of the peak HR achieved during the initial incremental test. Participants will be encouraged to breathe normally and avoid the Valsalva maneuver.
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Other: Isometric exercise — In each arm, participants will execute an isometric exercise, in which they will perform 4 repetitions of 2 minutes.
  Arms: Isometric Handgrip Session; Isometric Wall Squat Session

SUMMARY:
Hypertension remains the main preventable cause of cardiovascular disease (CVD) and all-cause mortality, both in Europe and globally. Resistant hypertension, a severe phenotype of hypertension, is defined as a blood pressure (BP) that remains above the management goal despite using three different antihypertensive agents of different classes at the maximum or maximum tolerated dose, or controlled BP on four or more antihypertensive medications. Hypertension remains a poorly controlled risk factor on a global scale and the prevalence of resistant hypertension is also growing - it is now estimated to be around 10-20%.

At the moment, there is robust evidence establishing the antihypertensive effects of exercise. The acute reduction of BP after a single bout of exercise is known as post-exercise hypotension.

In recent years, the number of investigations into the benefits of isometric exercise in the treatment of hypertension has increased, due to its ease of access and potential for use. In a recently published meta-analysis, the authors pointed to isometric exercise as the most effective type of exercise in reducing systolic and diastolic BP.

Given the scarceness of data regarding the safety and efficacy of isometric exercise in individuals with resistant hypertension and since the acute response to exercise may help to identify people who respond to exercise as antihypertensive therapy, the objective of this study is to analyse the acute effect on BP levels of two different isometric exercises - isometric handgrip (IHG) and isometric wall squat (IWS), regarding safety and efficacy, in people with resistant hypertension.

The aim is to analyse if isometric exercises are safe in this population, through the assessment of BP during the execution of the exercises. Besides that, the comparison of IHG and IWS with the control session and between one and another, will help to understand which form of isometric exercise is most effective and has the longest lasting impact on reducing BP.

Each participant must complete an acclimatization session, in which the procedures will be explained, data will be collected and the intensity of IHG and IWS will be assessed. Subsequently, each participant must complete three randomly assigned experimental sessions: a non-exercise control session and two exercise sessions, in which they will follow the protocols currently used in the literature (IHG at 30% of Maximum Voluntary Contraction and IWS at 95% of peak Heart Rate).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 75 years old, previously diagnosed with resistant hypertension, and on stable medication for at least 6 months.

Exclusion Criteria:

* People with secondary hypertension, heart failure, peripheral artery disease, atrial fibrillation, chronic obstructive pulmonary disease or renal failure; people with a cerebro-cardiovascular event in the previous 3 months; people with changes in pharmacological therapy in the previous 6 months; trained people (with regular participation (≥ 2x/week) in exercise training programs in the previous 3 months); people who have any contraindication to exercise; people with neurological and/ or orthopaedic conditions that will interfere with their participation in exercise, such as Parkinson's disease or knee osteoarthritis. Participants with low score (<6) on the MMAS-8 will also be excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | Blood Pressure (in mmHg) will be assessed 15 minutes after the intervention and then every 20 minutes after each intervention session (exercise sessions and control session) until 12 hours after session
  Change from baseline values of Ambulatory Systolic and Dyastolic Blood Pressure Monitoring (in mmHg)

SECONDARY OUTCOMES:
Office Blood Pressure | Systolic and Dyastolic BP will be measured immediately before the intervention session, during the exercise sessions (at 30 seconds and 90 seconds of each repetition of the handgrip and the wall squat) and 15 minutes after each intervention session
  Systolic and Dyastolic blood pressure (in mmHg) will be measured using automatic oscillometric (change from baseline will be calculated)
Adverse Events | Adverse events that occur during the intervention sessions, immediately after the intervention sessions or until 48 hours after the exercise sessions will be recorded
  Number and severity of adverse events that occur during or after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Ribeiro, PhD, Study Chair — University of Aveiro; Linda Pescatello, PhD, Study Chair — University of Connecticut; Ana Rita Pereira, MD, Study Chair — Local Health Unit of the Aveiro Region
Locations (1):
- Local Health Unit of the Aveiro Region, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of this article, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publication of the main results and up to five years.
Access Criteria: Individual participant data will be available for researchers who provide a methodologically sound proposal (e.g. individual participant meta-analysis).